CLINICAL TRIAL: NCT03124030
Title: Evaluation of the Intra- and Post- Operative Bleeding After Simple Dental Extraction in Direct Oral Anticoagulant Therapy Patients: a Longitudinal Observational Cohort Study
Brief Title: Intra- and Post- Operative Bleeding After Simple Dental Extraction in Direct Oral Anticoagulant Therapy
Acronym: NOADB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, prof. Roberto Di Lenarda, Prof., University of Trieste
Other Study IDs: NOADB_extractive
Record Dates: First submitted 2017-03-30; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Anticoagulant-induced Bleeding; Dental Diseases
Keywords: direct oral anticoagulant; oral anticoagulant therapy; dental extraction; bleeding complication; atrial fibrillation; deep venous thrombosis
MeSH Terms: conditions — Stomatognathic Diseases; Atrial Fibrillation; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Direct Oral Anticoagulants: assuming Pradaxa or Apixaban or Eliquis; undergo simple dental extraction
  Interventions: Procedure: simple dental extraction
- Oral Anticoagulant therapy: assuming Coumadin or Sintrom; undergo simple dental extraction
  Interventions: Procedure: simple dental extraction

INTERVENTIONS:
Procedure: simple dental extraction — dental extraction is performed by an expert oral surgeon within 20 minutes. Non-resorbable suture are applied
  Other Names: surgical dental avulsion

SUMMARY:
Direct Oral Anticoagulants were recently approved for medical treatment of several condition such as, non valvular atrial fibrillation, deep venous thrombosis, and others, substituting sometimes the conventional oral anticoagulants. The aim of the present study is to observe the possible difference in intra-operative and post-operative bleeding events for single dental extraction.

DETAILED DESCRIPTION:
Many protocols of drug suspension for surgical procedure has been designed, since the introduction of anticoagulant or antiplatelet medications. Nowadays it is not certain if suspension could give more costs than benefits for the surgical procedure itself. With the recent development of the Direct Oral Anticoagulant it is still unclear whether these medications might bring more bleeding events in the intra-operative and post-operative phase after oral surgery procedure, equal to, or more than Oral Anticoagulant Therapy. The purpose of this study is to assess the degree of intra- and post-operative bleeding complication between direct oral anticoagulant therapy patients and Oral Anticoagulant Therapy patients.

ELIGIBILITY:
Direct Oral Anticoagulant

Inclusion Criteria:

1. Male and female patients at 20 or more years of age.
2. Healthy patients (≤ American Society of Anesthesiologists 3).
3. Regular oral anticoagulant therapy assumed from at least 3 months with the following molecula: Dabigatran (PRADAXA), Rivaroxaban (XARELTO), Apixaban (ELIQUIS), Edoxaban (LIXIANA).
4. Indication for extraction of a single tooth.
5. No other contraindications for tooth extraction.
6. Accepted platelet count within 7 days prior to the procedure has to be > 50000 mg/dl.
7. Signed informed consent.

Exclusion Criteria:

1. Smoke > 10 cigarettes per day.
2. Assumption of any antiplatelet medication.
3. Assumption of Heparin medication.
4. Assumption of oral anticoagulant medications (Warfarin, Coumadin).
5. Wash-out period after antiplatelet or Heparin medication at least 15 days.
6. Assumption of food or drugs that may alter direct oral anticoagulant blood values.
7. Uncontrolled Hypertension.
8. Uncontrolled Diabetes
9. Chronic Hepatitis and/or reduction of hepatic function
10. Coagulopathy (in excess of defect)
11. Anamnestically known intolerance to one of the drugs applied or to their ingredients or to drugs of similar chemical structure.
12. Head and neck radiotherapy (previous 10 years).
13. Chemotherapy (previous 2 years).
14. Participation of the patient in another clinical trial within the last four weeks before enrollment in this trial.
15. Incapability of assessing essence and possible consequences of the trial (e.g. alcoholism).
16. Pregnant or breastfeeding women.
17. Evidence suggesting that the patient is not likely to follow the study protocol (e.g. lack of compliance).

Oral Anticoagulant Therapy

Inclusion Criteria:

1. Male and female patients at 20 or more years of age.
2. General health status (< American society of anesthesiologist a 3).
3. Regular oral anticoagulant therapy assumed from at least 3 months with the following molecula: Warfarin (COUMADIN), acenocoumarol (SINTROM).
4. Indication for extraction of a single tooth.
5. No contraindications for tooth extraction.
6. Accepted platelet count within 7 days prior to the procedure has to be > 50000 mg/dl.
7. International Normalized Ratio measured within 7 days prior to the procedure should between 2.0 and 3.0.
8. No diet changes within the week before blood sampling (avoiding interacting food)
9. Signed informed consent.

Exclusion Criteria:

1. Smoke > 10 cigarettes per day.
2. Assumption of any antiplatelet medication.
3. Assumption of any Heparin medication.
4. Assumption of any direct oral anticoagulant medication.
5. Uncontrolled Hypertension.
6. Uncontrolled Diabetes.
7. Chronic Hepatitis and/or reduction of hepatic function
8. Coagulopathy (in excess of defect)
9. Wash-out period after antiplatelet or Heparin medication at least 15 days.
10. Anamnestically known intolerance to one of the drugs applied or to their ingredients or to drugs of similar chemical structure.
11. Assumption of food or drugs that may alter oral anticoagulant blood values.
12. Head and neck radiotherapy (previous 10 years).
13. Chemotherapy (previous 10 years).
14. Participation of the patient in another clinical trial within the last four weeks before enrollment in this trial.
15. Incapability of assessing essence and possible consequences of the trial (e.g. alcoholism).
16. Pregnant or breastfeeding women.
17. Evidence suggesting that the patient is not likely to follow the study protocol (e.g. lack of compliance).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiovascular patient assuming oral anticoagulant therapy (conventional or direct)
Sampling Method: Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-11-15 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
post-operative bleeding complication | 30 minutes
  questionnaire is provided to the patient for bleeding characterization

SECONDARY OUTCOMES:
oral health status | 1 week before
  examination of the oral cavity, registration of periodontal indices
cardiological assessment | 1 week before
  registration of the Atrial Fibrillation Stroke Risk score
bleeding risk assessment | 1 week before
  registration of the Score for Major Bleeding Risk score
intra-operative bleeding | intra-operative
  a standardized cotton roll is weighted after imbibition on the post-extractive alveolus for 20 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Fulvia Costantinides, Dr., Study Chair — University of Trieste; Federico Berton, Dr., Study Director — University of Trieste; Roberto Di Lenarda, Prof., Principal Investigator — University of Trieste; Erika Visintini, Dr., Study Chair — University of Trieste
Locations (1):
- Clinica Odontoiatrica e Stomatologica, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: a discussion paper on clinical implications of oral anticoagulants — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4731944/